CLINICAL TRIAL: NCT00799721
Title: Urine VEGF Levels in Very Low Birth Weight (VLBW) Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Anke Reinhold, Charité University Berlin
Other Study IDs: EA2/072/08-1
Record Dates: First submitted 2008-11-28; First posted 2008-12-01 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-08

CONDITIONS: Infant, Very Low Birth Weight
Keywords: ROP; VLBW; Epo; IUGR; VEGF; sFLT-1; very low birth weight infants; retinopathy of prematurity; erythropoietin therapy and risk of ROP
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples that are centrifugated to get rid of any cells where stored at -80°C until ELISA is done.

GROUPS / COHORTS (2):
- 1: VLBW infants with erythropoietin therapy
- 2: VLBW infants without erythropoietin therapy.

SUMMARY:
VLBW infants are at risk of developing retinopathy of prematurity (ROP). In the first phase of ROP there is a down-regulation of retinal VEGF-expression because of postnatal relative hyperoxia, followed by an upregulation of VEGF mediated through retinal hypoxia, which leads to pathologic vessel formation. VEGF acts through binding to the specific receptor FLT-1, the soluble form sFLT-1 is a specific antagonist of VEGF action. Erythropoietin, given to VLBW infants to prevent anemia, may stimulate VEGF-production in neuronal cells. Currently, there are no data published about VEGF urine-levels in VLBW infants and it is not known, if urine VEGF-levels may serve as a non-invasive marker of ROP-risk. Further shall be investigated, if erythropoietin-therapy increases urine VEGF-levels and if there is a correlation with ROP-development.

ELIGIBILITY:
Inclusion Criteria:

* gestational age < 32 weeks
* birth weight <1500g

Exclusion Criteria:

* absent written consent by parents
* connatal eye malformation

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pretarem infants of less than 32 weeks of gestation or birth weight below 1500g.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-02 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Development of ROP | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Virchow-Hospital, Berlin, State of Berlin, Germany